CLINICAL TRIAL: NCT04166877
Title: Magnesium Infusion for Pain Management in Critically Ill Trauma Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1440730
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Trauma; Acute Pain
Keywords: magnesium sulfate; trauma; acute pain
MeSH Terms: conditions — Wounds and Injuries; Acute Pain | interventions — Magnesium Sulfate; Injections

STUDY DESIGN:
Intervention Model Description: Single center, investigator-initiated, randomized, double-blinded, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Group (Experimental): The magnesium group arm will receive a 40 mg/kg IBW (maximum 4 g) bolus of intravenous magnesium sulfate, followed by a continuous infusion of 0.5 g/hr for a total of 24 hours.
  Interventions: Drug: Magnesium Sulfate in Parenteral Dosage Form
- Control Group (Placebo Comparator): The control arm will receive the same volume and rate of saline as if they were in the experimental group.
  Interventions: Drug: Normal saline placebo

INTERVENTIONS:
Drug: Magnesium Sulfate in Parenteral Dosage Form — IV bolus followed by continuous infusion for 24 hours
  Arms: Magnesium Group
Drug: Normal saline placebo — IV bolus followed by continuous infusion for 24 hours
  Arms: Control Group

SUMMARY:
Magnesium is a naturally occurring mineral that is important for your body and brain. Magnesium sulfate (study drug) is a medication containing magnesium that is commonly used to improve low blood levels of magnesium. Magnesium sulfate has also proven to be successful in managing pain before and after surgery. However, this drug has primarily been used for pain control in patients undergoing surgery. Patients in the ICU with injuries also need good pain control. Using magnesium may assist in decreasing narcotic (pain reliever) requirements and provide another non-narcotic drug for pain control.

The purpose of this study is to test the effectiveness of continuous, intravenous (into or within a vein using a needle) administration of magnesium sulfate for pain control in trauma patients admitted to the adult Intensive Care Unit. This will be compared to intravenous normal saline (salt solution).

DETAILED DESCRIPTION:
This is a single center, double blind, randomized controlled study to demonstrate the effectiveness of continuous, intravenous administration of magnesium sulfate as compared to placebo in decreasing pain in critically injured patients.

Study Hypothesis The primary hypothesis is that continuous infusion magnesium sulfate will significantly decrease opioid requirements and pain scores in critically ill patients.

Background Magnesium is one of the most abundant cations in the human body. The physiologically active form of magnesium, ionized magnesium, is involved in hundreds of enzyme reactions that are important for homeostasis, action potentials, and membrane stability, among others.[Seo, et al] Hypomagnesemia is one of the most common electrolyte disturbances in the hospitalized patient, especially in the critically ill population. Studies have established that low magnesium levels increase mortality and morbidity in the critically ill patient,[Upala, et al] and thus magnesium is often repleted with intermittent infusion. Outside of its role in enzyme reactions, magnesium was discovered to have analgesic effects approximately twenty years ago.[Albrecht, et al] It appears to potentiate morphine analgesia, attenuate morphine tolerance, and suppress neuropathic pain.[Albrecht, et al] At a mechanistic level, these effects are thought to be secondary to magnesium regulating calcium influx into cells and antagonizing NMDA receptors in the central nervous system.

Magnesium has long been utilized in prevention and management of preeclampsia and eclampsia. A typical dosing regimen in this setting involves a 4 g loading dose of magnesium sulfate, followed by a magnesium infusion of 1-2 g/hr. When compared to eclampsia regimens, studies investigating the role of magnesium sulfate in multimodal surgical pain management consistently use lower doses. Even with this dosing, multiple trials have shown reduced postoperative pain and analgesic requirements.[Albrecht, et al, Sousa, et al, Hwang, et al, Shariat, et al] In one example, Shariat Moharari and others used a regimen of 40 mg/kg magnesium bolus followed by 10 mg/kg/hr infusion in perioperative gastrointestinal surgery patients, without adverse effects.[Shariat, et al]

Normal reference range for serum magnesium has been defined as approximately 0.7-1 mmol/L (1.5-2 mEq/L or 1.7-2.4 mg/dL).[Williamson, et al] Tramer et al. reported that a 3 g bolus dose of magnesium sulfate followed with 0.5 g/hr infusion for 20 hours resulted in an increase from baseline serum magnesium of approximately 0.6 mmol/L. Despite the higher post-treatment serum magnesium levels in the treatment group, no difference in safety outcomes was noted in comparison to the control group receiving 0.9% sodium chloride.[Tramer,et al] Similarly, Ozcan et al. found that 30 mg/kg bolus dose of magnesium sulfate followed by infusion of 10 mg/Kg/hr for 48 hours resulted in an increased serum magnesium level from baseline by approximately 0.7 mmol/L. The noted increase in serum magnesium level in this study also did not translate into any difference in safety endpoints between the intervention group and control group receiving 0.9% sodium chloride.[Ozcan, et al] Initial signs of magnesium toxicity following administration of magnesium sulfate have been reported to occur at serum magnesium levels greater than 3.5-5 mmol/L.[Lu, et al, Jahnen-Dechent, et al]

Despite the successful use of magnesium in perioperative pain management, it has yet to be applied in patient populations outside of the operating room. Given the need for adequate pain control among critically ill patients with traumatic injuries, the use of magnesium for pain management may assist in decreasing opioid requirements and provide another non-opioid adjunct for pain control.

Methods:

All trauma patients admitted to an adult ICU are screened during the first 24 hours after admission. If they meet criteria for admission to the study, an informed consent will be obtained. Patients meeting eligibility will be randomized by the Investigational Drug Service in a computer-generated, blinded block, 1:1 ratio to treatment with either magnesium sulfate (diluted appropriately in normal saline per standard procedures) or placebo (normal saline)."

Opioid administration will be recorded per usual nursing protocol in the electronic medial record. Heart rate, mean arterial pressure (MAP), respiratory rate, and RASS will be recorded at least every two hours per unit protocol.

A study worksheet will be posted at bedside for consistent collection of pain scores and CAM. Pain will be assessed per unit protocol using the numeric rating scale, with zero representing no pain and ten representing the worst pain imaginable.

The EMR will be reviewed; opioid administration, pain scores, and vital signs will be transferred to a separate data sheet through REDCap (Research Electronic Data Capture) software.

The primary outcome measure will be the total opioid requirement during the 24 hours of magnesium infusion. We performed this power analysis based on a recent retrospective cohort study performed at our institution.[Hamrick, et al] We estimate that the 24 hour OME requirement will decrease from 70 mg in the control group to 50 mg in the treatment group, with a standard deviation of 50 mg in each group, leading to an effect size of 0.4. Using the statistical program G*Power 3.0.1 with an effect size of 0.4, alpha of 0.05, power of 0.8, and equal allocation ratios, a sample size of 78 patients per group would be required.

Data will be assessed for normality by assessing distribution skewness and kurtosis. Depending on these results, t-tests or Wilcoxon rank-sum tests for two groups will be used to assess the primary outcome of total opioid dose. Other data, including pain scores, that is collected repeatedly will be analyzed with two-way repeated measures analysis of variance, with subsequent pair-wise comparison for any significant findings. Statistical significance will be set at a P value of less than 0.05. We will use SAS to perform the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients admitted to an adult intensive care unit
* Signed informed consent
* Hospital or trauma multimodal pain management order set used for pain management
* Ages 18-99

Exclusion Criteria:

* Admission to the Pediatric Intensive Care Unit.
* Head Abbreviated Injury Score (AIS) of greater than 1
* Known heart failure with reduced ejection fraction (EF < 40%)
* Renal failure (GFR < 60)
* Cardiac arrhythmia (except for sinus tachycardia)
* Greater than 5% TBSA burn injuries
* Moderate to severe alcohol withdrawal protocol ordered for patient
* Regular use of opioids in the week prior to injury
* Receiving continuous infusion of opioids
* Patients expected to require general anesthesia between 24 and 48 hours after admission (during study drug administration)
* Patients unable to provide consent is unavailable
* Patients unable to provide a pain score
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2019-12-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
total opioid requirements during study drug infusion | 24 hours during study drug infusion
  oral morphine equivalents, OME

SECONDARY OUTCOMES:
pain scores | daily x 4 days
  numeric pain rating scale as reported by patient
Total oral morphine equivalents | daily x 4 days
ICU length of stay | through the patient's hospitalization for this injury, an average of 10 days
ICU-free days | 14 days
  14 days minus the number of ICU days
Hospital length of stay | through the patient's hospitalization for this injury, an average of 10 days
Development of bradycardia | 24 hours during study drug infusion
Development of other dysrhythmia | 24 hours during study drug infusion
Respiratory depression | 24 hours during study drug infusion
  Episodes of respiratory depression as measured by a respiratory rate less than 8
Prevalence of Richmond Agitation-Sedation Scale of -3 to -5 | 24 hours during study drug infusion
  Episodes of a -3 to -5 Richmond Agitation-Sedation Scale score

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seo JW, Park TJ. Magnesium metabolism. Electrolyte Blood Press. 2008 Dec;6(2):86-95. doi: 10.5049/EBP.2008.6.2.86. Epub 2008 Dec 31. PMID 24459527
- [Background] Upala S, Jaruvongvanich V, Wijarnpreecha K, Sanguankeo A. Hypomagnesemia and mortality in patients admitted to intensive care unit: a systematic review and meta-analysis. QJM. 2016 Jul;109(7):453-459. doi: 10.1093/qjmed/hcw048. Epub 2016 Mar 24. PMID 27016536
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] Sousa AM, Rosado GM, Neto Jde S, Guimaraes GM, Ashmawi HA. Magnesium sulfate improves postoperative analgesia in laparoscopic gynecologic surgeries: a double-blind randomized controlled trial. J Clin Anesth. 2016 Nov;34:379-84. doi: 10.1016/j.jclinane.2016.05.006. Epub 2016 Jun 5. PMID 27687417
- [Background] Hwang JY, Na HS, Jeon YT, Ro YJ, Kim CS, Do SH. I.V. infusion of magnesium sulphate during spinal anaesthesia improves postoperative analgesia. Br J Anaesth. 2010 Jan;104(1):89-93. doi: 10.1093/bja/aep334. PMID 19933175
- [Background] Shariat Moharari R, Motalebi M, Najafi A, Zamani MM, Imani F, Etezadi F, Pourfakhr P, Khajavi MR. Magnesium Can Decrease Postoperative Physiological Ileus and Postoperative Pain in Major non Laparoscopic Gastrointestinal Surgeries: A Randomized Controlled Trial. Anesth Pain Med. 2013 Dec 6;4(1):e12750. doi: 10.5812/aapm.12750. eCollection 2014 Feb. PMID 24660146
- [Background] Hamrick KL, Beyer CA, Lee JA, Cocanour CS, Duby JJ. Multimodal Analgesia and Opioid Use in Critically Ill Trauma Patients. J Am Coll Surg. 2019 May;228(5):769-775.e1. doi: 10.1016/j.jamcollsurg.2019.01.020. Epub 2019 Feb 21. PMID 30797081
- [Background] Williamson M. A., Snyder L. M., Wallach J. B. Wallach's Interpretation of Diagnostic Tests. 9th. Philadelphia, PA, USA: Wolters Kluwer/Lippincott Williams & Wilkins; 2011. xvi, 1143.
- [Background] Tramer MR, Schneider J, Marti RA, Rifat K. Role of magnesium sulfate in postoperative analgesia. Anesthesiology. 1996 Feb;84(2):340-7. doi: 10.1097/00000542-199602000-00011. PMID 8602664
- [Background] Ozcan PE, Tugrul S, Senturk NM, Uludag E, Cakar N, Telci L, Esen F. Role of magnesium sulfate in postoperative pain management for patients undergoing thoracotomy. J Cardiothorac Vasc Anesth. 2007 Dec;21(6):827-31. doi: 10.1053/j.jvca.2006.11.013. Epub 2007 Feb 7. PMID 18068060
- [Background] Lu JF, Nightingale CH. Magnesium sulfate in eclampsia and pre-eclampsia: pharmacokinetic principles. Clin Pharmacokinet. 2000 Apr;38(4):305-14. doi: 10.2165/00003088-200038040-00002. PMID 10803454
- [Background] Jahnen-Dechent W, Ketteler M. Magnesium basics. Clin Kidney J. 2012 Feb;5(Suppl 1):i3-i14. doi: 10.1093/ndtplus/sfr163. PMID 26069819